CLINICAL TRIAL: NCT05879783
Title: Use of Probe-based Confocal Laser Endomicroscopy to Perform Optical Biopsy for Peritoneal Nodules in Colorectal Cancer Patients During Surgery
Brief Title: Optical Biopsy for Peritoneal Nodules in Colorectal Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2023-088
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Confocal laser endomicroscopy; Optical biopsy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probe-based confocal laser endomicroscopy biopsy (Experimental): In this study , pCLE-based optical biopsy will be successively performed for peritoneal nodules in colorectal cancer patients during surgical operation.
  Interventions: Diagnostic Test: Confocal laser endomicroscopy

INTERVENTIONS:
Diagnostic Test: Confocal laser endomicroscopy — After intravenous injection of fluorescein sodium, pCLE-based optical biopsy will be performed.

SUMMARY:
During surgery, peritoneal metastasis is typically confirmed pathologically through resection sample. However, this process can be time-consuming when utilizing intro-operative frozen section pathology. To address this issue, we propose utilizing confocal laser endomicroscopy to provide in situ, real-time, and in-vivo diagnosis of suspected peritoneal nodules as cancer metastasis during surgery.

DETAILED DESCRIPTION:
Peritoneal metastasis is a common metastatic site in colorectal cancer patients, and those with peritoneal metastasis often have a poor prognosis. During surgery, peritoneal metastasis is confirmed pathologically through resection sample, but frozen section pathology can take up to 30 minutes, which is a significant amount of time.

To address this issue, we suggest utilizing probed-based confocal laser endoscopy (pCLE), a novel endoscopic adjunct that enables real-time in vivo histological examination of mucosal surfaces. By using intravenous fluorescent agents, pCLE highlights certain mucosal elements that facilitate an optical biopsy in real time.

By providing a promising optical biopsy, CLE has the potential to enable in situ, real-time, and in vivo diagnosis of colorectal cancer patients with peritoneal nodules during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age from over 18 to under 85 years
2. American Society of Anesthesiology (ASA) score class I,II,or III
3. Colorectal cancer
4. Patients who be about to undergo surgical treatment
5. Written informed consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Acute renal insufficiency or stage II to IV chronic renal insufficiency
3. Patients with severe liver damage
4. Asthma patients or patients with allergic constitution

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of pCLE optical biopsy | 7 days
  The investigators will use pCLE optical biopsy for peritoneal nodules in colorectal cancer patients and compare the pathological diagnosis between optical biopsy and surgically resected specimens.

SECONDARY OUTCOMES:
Sensitivity, specificity of pCLE optical biopsy | 7 days
  The investigators will use pCLE optical biopsy for peritoneal nodules in colorectal cancer patients and compare the pathological diagnosis between optical biopsy and surgically resected specimens.
The positive predictive value and negative predictive value of pCLE optical biopsy | 7 days
  The investigators will use pCLE optical biopsy for peritoneal nodules in colorectal cancer patients and compare the pathological diagnosis between optical biopsy and surgically resected specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D., Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mansour MR, Caycedo-Marulanda A, Davis BR, Alawashez A, Docimo S, Qureshi A, Tsuda S. SAGES TAVAC safety and efficacy analysis confocal laser endomicroscopy. Surg Endosc. 2021 May;35(5):2091-2103. doi: 10.1007/s00464-020-07607-3. Epub 2020 May 13. PMID 32405892
- [Background] Baratti D, Kusamura S, Pietrantonio F, Guaglio M, Niger M, Deraco M. Progress in treatments for colorectal cancer peritoneal metastases during the years 2010-2015. A systematic review. Crit Rev Oncol Hematol. 2016 Apr;100:209-22. doi: 10.1016/j.critrevonc.2016.01.017. Epub 2016 Jan 22. PMID 26867984